CLINICAL TRIAL: NCT07058922
Title: Acute Effects of Powdered Beetroot Extract Supplementation on the Microcirculation of Resistant Hypertensive Individuals
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Institute of Cardiology, Laranjeiras, Brazil (Other Government)
Responsible Party: Principal Investigator, Eduardo Tibirica, MD, PhD, senior researcher, National Institute of Cardiology, Laranjeiras, Brazil
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAAE70847523.9.0000.5272
Record Dates: First submitted 2025-07-01; First posted 2025-07-10 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Resistant Arterial Hypertension
Keywords: arterial hypertension; systemic microcirculation; beetroot extract
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Nutritional supplement containing a powdered beetroot extract - 400 mg of nitrate per dose will be used in the supplement group, administered orally at a daily amount of 10 g.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- beetroot powder extract supplement (Experimental): A powdered beetroot extract supplement containing 400 mg of nitrate per dose will be used in the supplement group, administered orally at a daily amount of 10 g.
  Interventions: Diagnostic Test: evaluation of systemic microvascular reactivity; Diagnostic Test: ABPM; Dietary Supplement: beetroot supplement
- placebo control (Placebo Comparator): An isocaloric, colored, and flavored supplement composed of maltodextrin will be orally administered.
  Interventions: Diagnostic Test: evaluation of systemic microvascular reactivity; Diagnostic Test: ABPM

INTERVENTIONS:
Diagnostic Test: evaluation of systemic microvascular reactivity — Evaluation of systemic microvascular reactivity using laser speckle contrast imaging.
Diagnostic Test: ABPM — Ambulatory blood pressure measuring: systolic, diastolic and mean arterial pressures
Dietary Supplement: beetroot supplement — A powdered beetroot extract supplement containing 400 mg of nitrate per dose will be used in the supplement group, administered orally at a daily amount of 10 g.
  Arms: beetroot powder extract supplement

SUMMARY:
Arterial hypertension is a major public health issue and is considered to be a new epidemic due to its high mortality and morbidity rates. Elevated blood pressure levels increase the risk of coronary artery disease, heart failure, stroke, chronic kidney disease and death. Dietary nitrate supplementation in the form of beetroot powder extract may offer a more accessible way to increase systemic nitric oxide availability and consequently promote vasodilation in these patients. However, studies are needed to assess its benefits in patients with hypertension.

DETAILED DESCRIPTION:
Methods and Analyses: This is a double-blind, placebo-controlled clinical trial in which patients with hypertension will be randomly assigned to two groups to receive either nitrate powder supplementation or placebo for a duration of 60 days. The primary outcome will be the reduction in blood pressure levels. Secondary outcomes will include systemic microvascular reactivity and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Resistant hypertensive patients, with a diagnosis documented in medical records, without any change in medication or increase in dosage in the past 30 days.

Exclusion Criteria:

* Patients will be excluded from the study if they have: neoplasms, heart failure, are using medications containing nitrate in their formulation, or have undergone renal denervation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Blood pressure | 60 days of tratment
  ABPM - measurement of systolic, diastolic and mean arterial pressure.

SECONDARY OUTCOMES:
Systemic microvascular reactivity | 60 days treatment

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Cardiology, Rio de Janeiro, Rio de Janeiro, Brazil